CLINICAL TRIAL: NCT05997329
Title: Nutrition Throughout the Treatment Course - Expanding Care From Hospital to Home
Acronym: NUTREAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); University of South-Eastern Norway (Other)
Responsible Party: Principal Investigator, Christine Henriksen, Associate professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 569956
Record Dates: First submitted 2023-06-26; First posted 2023-08-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Amyloid; Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyFood (App for diet record) (Experimental): Use of an App for diet record
  Interventions: Other: App for diet record (MyFood)
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: App for diet record (MyFood) — Patients in the intervention group will record their food intake, tube feeding, nutrition-related symptoms and body weight in the MyFood app in at least three consecutive days in advance of follow-up.The patients will thus be able to keep track of their nutrition status. They will also have access to nutrition tips for how to reach requirements if they struggle to eat sufficiently or relief symptoms that can affect food intake.Healthcare staff at the hospital and outpatient clinics will use MyFood to monitor the patient's nutrition and document this information in the electronic patient record. They will also receive decision support tailored to each individual patient, e.g. recommendations for how to use oral nutrition supplements if the patient's intake of energy or protein is too low. Patients who struggle to fulfill their requirements will receive an additional referral to a registered dietitian for nutrition treatment between week 5 and 11.
  Arms: MyFood (App for diet record)

SUMMARY:
Patients with cancer have increased risk of malnutrition due to the disease itself and the treatment regimen they undergo. This is particularly relevant for patients with head and neck cancer (HNC), where 74%-95% are malnourished. HNC is a heterogenous group of cancers, including oral cavity, larynx, pharynx and salivary glands. The present project will study the effectiveness and implementation of remote patient monitoring of nutrition and tailored nutrition support throughout the treatment course in patients with head and neck cancer. The implementation will be evaluated in a randomized controlled trial (RCT), and the aim of the project is to reduce the prevalence of malnutrition and increase the quality of life among patients with HNC.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer
* Older than 18 years

Exclusion Criteria:

* Patients admitted with the classification of malignant tumors (TNM) stage 4
* Terminal condition (life expectancy < 6 months)
* Patients who do not understand the Norwegian language.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Malnutrition_PGSGA | 18 weeks
  Measured by the: Patient-Generated Subjective Global Assessment (PG-SGA). The tool categories participants into: category A (Well-nourished), B (Moderately malnutrition or possible malnutrition), or C (serious malnutrition)

SECONDARY OUTCOMES:
Malnutrition GLIM | 18 weeks
  Malnutrition measured by the objective method developed by the Global Leadership Initiative on Malnutrition (GLIM). The GLIM-criteria also categories the participants i three groups: Well-nourished, moderate malnutrition and severe malnutrition.
Weight change | 18 weeks
  weight measurements
Nutrition intake | 18 weeks
  24-hour recall interviews
Body composition | 18 weeks
  Bioelectrical Impedance Analysis (BIA)
Health-related quality of life | 18 weeks
  EuroQol Research Foundation, Netherlands (EQ5D-5L). Assess health in 5 dimensions each of which has three response levels (1: No problems, 2: some problems and 3: extreme problems/unable to do).
Number of Participants compliant to the intervention | 18 weeks
  Review of reported use of the MyFood app in the electronic patient record
Number of patients with non-elective readmissions | 18 weeks
  Review of readmissions in the electronic patient record

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - University of Oslo, Oslo, Oslo County
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Severinsen F, Varsi C, Andersen LF, Henriksen C, Paulsen MM. Experiences with nutritional follow-up and barriers and opportunities of implementing digital seamless nutrition care in the head and neck cancer treatment course: a qualitative study from patient, family caregiver, and healthcare professional perspectives. BMC Health Serv Res. 2025 Oct 14;25(1):1358. doi: 10.1186/s12913-025-13542-7. PMID 41088125